CLINICAL TRIAL: NCT06445673
Title: A Prospective, Multicenter, International Non-interventional, Observational Cohort Study to Observe Long-term Treatment Patterns and Real-word Outcomes in PAH Group I Patients Previously Participating in TripleTRE - TripleTRE-NIS
Brief Title: A Prospective Non-interventional Observational Study to Observe Long-term Treatment and Outcomes in Pulmonary Arterial Hypertension (PAH) Patients
Acronym: TripleTRE-NIS
Status: Enrolling by invitation | Type: Observational
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Other Study IDs: TREV1-10P.NIS
Record Dates: First submitted 2024-05-29; First posted 2024-06-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TripleTRE NIS patients: all patients previously treated within the TripleTRE trial who are willing to participate in this NIS

SUMMARY:
The goal of this observational study is to learn about the long-term development and outcomes of different treatment patterns of patients who initially participated in the TripleTRE study.

The primary objective of this non-interventional follow-up study is to assess the long-term real-world clinical outcomes, including disease progression and survival rates, in patients who initially participated in and completed the randomized TripleTRE trial.

Planned observation duration per patient is a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients previously participating in the randomized TripleTRE trial who are able and willing to provide a signed informed consent for study participation in NIS

Exclusion Criteria:

1. Lost to follow-up patients of TripleTRE study
2. Patients who discontinued all medicinal PAH treatments (e.g. after successful lung transplantation)
3. Patients who withdrew from the initial TripleTRE trial due to significant non-compliance with trial requirements (not adhering to therapy, not coming to hospital visits)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who participated in the TripleTRE study and who have not been lost to follow-up and have given a written informed consent for their participation in the NIS.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Time to death or lung transplantation | up to year 3
Time to first clinical worsening | up to year 3
  clinical worsening is defined as fulfilling on of the following criteria:
  * PAH related death (including all deaths where PAH cannot be excluded as cause)
  * Lung transplantation due to PAH
  * PAH-related hospitalization
  * Post baseline decrease in 6MWD by 15%
  * Post baseline worsening of WHO FC
Total number of clinical worsenings | up to year 3
  clinical worsening is defined as fulfilling on of the following criteria:
  * PAH related death (including all deaths where PAH cannot be excluded as cause)
  * Lung transplantation due to PAH
  * PH-related hospitalization
  * Post baseline decrease in 6MWD by 15%
  * Post baseline worsening of WHO FC

SECONDARY OUTCOMES:
Long-term change in 6MWD | up to year 3
  6-Minute Walking Distance (6MWD) will be measured in meters
Long-term change in PAH treatment regimens | up to year 3
  any change or addition of new PH medication including dosing in time
Long-term change in risk status | up to year 3
  Risk status measured by simplified four-strata risk-assessment tool
Long-term change in WHO FC | up to year 3
  World Health Organization Functional Class (WHO FC) is categorized from I (no symptoms) to IV (severe dyspnea and symptoms)
Long-term change in BDS | up to year 3
  BDS - Borg Dyspnea Score, ranging from 0 (no exertion) to 10 (maximum)
Long-term change in NT-proBNP/BNP | up to year 3
  NT-proBNP/BNP: N-terminal pro Brain Natriuretic Peptide
Long-term change in Pulmonary Vascular Resistance (PVR) | up to year 3
  PVR to be measured in WU Parameter will be collected according to clinical routine
Long-term change in mean Pulmonary Arterial Pressure (mPAP) | up to year 3
  mPAP to be measured in mmHg Parameter will be collected according to clinical routine
Long-term change in Right Atrial Pressure (RAP) | up to year 3
  RAP to be measured in mmHg Parameter will be collected according to clinical routine
Long-term change in mean Right Atrial Pressure (mRAP) | up to year 3
  mean Right Atrial Pressure (mRAP) to be measured in mmHg Parameter will be collected according to clinical routine
Long-term change in Cardiac Index (CI) | up to year 3
  Cardiac index (CI) measured in liters per minute per square meter Parameter will be collected according to clinical routine
Long-term change in Cardiac Output (CO) | up to year 3
  Cardiac output (CO) measured in liters per minute Parameter will be collected according to clinical routine
Long-term change in Pulmonary capillary wedge pressure (PCWP) | up to year 3
  Pulmonary capillary wedge pressure (PCWP) measured in mmHg Parameter will be collected according to clinical routine
Long-term change in Stroke volume index (SVI) | up to year 3
  Parameter will be collected according to clinical routine
Long-term change in RV-PA coupling | up to year 3
  RV-PA coupling estimated by the ratio of tricuspid annular plane systolic excursion by pulmonary artery systolic pressure Parameter will be collected according to clinical routine
Long-term change in RV end-diastolic area (RVEDA) | up to year 3
  RV end-diastolic area (RVEDA) measured in square centimeters Parameter will be collected according to clinical routine
Long-term change in RV end-systolic area (RVESA) | up to year 3
  RV end-systolic area (RVESA) measured in square centimeters Parameter will be collected according to clinical routine
Long-term change in RV fractional area change (RVFAC) | up to year 3
  RV fractional area change (RVFAC) calculated in % Parameter will be collected according to clinical routine
Long-term change in Right Atrium (RA) area | up to year 3
  Right Atrium (RA) area in square centimeters Parameter will be collected according to clinical routine
Long-term change in Pericardial effusion | up to year 3
  Pericardial effusion assessment will be done and rated as yes/no Parameter will be collected according to clinical routine
Long-term change in Right ventricular ejection fraction (RVEF) | up to year 3
  Parameter will be collected according to clinical routine

OTHER OUTCOMES:
Frequency and seriousness of adverse events (AE) and adverse drug reactions (ADR) | up to year 3
  This includes:
  * Adverse events (S)AEs
  * Adverse drug reactions (S)ADRs related to any of PAH treatments
  * Adverse events related to underlying diagnosis, PAH
Long-term change in QoL using European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) questionnaire | up to year 3
  The EQ-5D-5L questionnaire consists of 2 parts - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale. The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. It should be noted that the numerals 1-5 have no arithmetic properties and should not be used as a cardinal score.
Long-term change in QoL using PAH-specific emPHasis-10 questionnaire | up to year 3
  Emphasis meaning something of special importance or significance. Please translate using the most appropriate term. The PH in emPHasis represents the condition Pulmonary Hypertension. The number 10 refers to the number of items in the questionnaire.
  This questionnaire is designed to determine how Pulmonary Hypertension (PH) affects patient's life. It refers to how PH affects or the impact that PH has on the patient's life.

CONTACTS AND LOCATIONS:
Locations (18):
- Austria (2):
  - Ordensklinikum Linz, Linz
  - Medical University Vienna, Vienna
- Czechia (2):
  - Fakultní Nemocnice Olomouc, Olomouc
  - Všeobecná fakultní nemocnice v Praze, Prague
- France (2):
  - Hôpital Bicêtre-- Assistance Publique Hopitaux de Paris, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (3):
  - DRK Kliniken Berlin Westend, Berlin
  - University Hospital Carl Gustav Carus of Technical University Dresden, Dresden
  - Universitätsmedizin Greifswald, Greifswald
- Hungary (2):
  - Gottsegen National Cardiovascular lnstitute, Budapest
  - Medical University of Szeged, Szeged
- Sapienza University of Rome, Rome, Italy
- Poland (2):
  - John Paul II Hospital Krakow, Krakow
  - Fryderyk Chopin Hospital in European Health Centre Otwock, Otwock
- Romania (2):
  - Emergency Institute for Cardiovascular Diseases Prof. Dr. C.C.Iliescu, Bucharest
  - Emergency Clinical County Hospital of Targu Mures, Târgu Mureş
- Spain (2):
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Ramon y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No